CLINICAL TRIAL: NCT06602752
Title: Impact Evaluation of the Global Alliance for Improved Nutrition (GAIN) Vegetables for All Program in Uganda
Brief Title: Vegetables for All Project in Uganda
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RTI International (Other)
Collaborators: Makerere University (Other)
Responsible Party: Principal Investigator, Valerie Flax, Senior Research Public Health Analyst, RTI International
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 424605
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Vegetable Consumption
Keywords: diet; vegetables; market intervention; social and behavior change communication intervention; bottom of pyramid; children; Uganda

STUDY DESIGN:
Intervention Model Description: Data will be collected through household surveys, vegetable vendor surveys, in-depth interviews, and focus group discussions. The study team has selected a subset of intervention FFZs for the evaluation and identified an equal number of geographic areas of similar size and level of urbanicity to serve as controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Active Comparator): The Vegetables for All project will create FFZs in low-income urban and peri-urban areas. FFZs are the last mile/point of purchase for delivering a variety of fresh, safe, and accessible vegetables to BoP households. The program will link vendors and farmers through market facilitators, support the uptake of digital solutions for vendors to access vegetables, and support district governments to improve market infrastructure. To encourage BoP parents of children 3-9 years to buy and consume more vegetables, the program will include a demand generation component.
  Interventions: Behavioral: Food system and demand generation
- Control/No Intervention (No Intervention): An equal number of geographic areas with similar levels of urban city to the intervention FFZs will serve as the control.

INTERVENTIONS:
Behavioral: Food system and demand generation — The Vegetables for All project will create FFZs in low-income urban and peri-urban areas. FFZs are the last mile/point of purchase for delivering a variety of fresh, safe, and accessible vegetables to BoP households. The program will link vendors and farmers through market facilitators, support the uptake of digital solutions for vendors to access vegetables, and support district governments to improve market infrastructure. To encourage BoP parents of children 3-9 years to buy and consume more vegetables, the program will include a demand generation component.
  Arms: Intervention

SUMMARY:
This study is an evaluation of the Global Alliance for Improved Nutrition (GAIN)'s Vegetables for All Project in Uganda. The aim of this program is to improve access to safe and fresh vegetables in FitFood Zones (FFZs) and generate demand for vegetables through a media campaign and FFZ branding. RTI and local partners will conduct impact and process evaluations of GAIN's program. The evaluation will include a mix of quantitative and qualitative methods and will be guided by the RE-AIM (reach, effectiveness, adoption, implementation, and maintenance) evaluation framework.

DETAILED DESCRIPTION:
Background: In Uganda, the goal of GAIN's 'Vegetables for All' project is to contribute to improving the dietary diversity of Ugandans through increased consumption of safe vegetables and greater use of vegetables in Ugandan cuisine, increasing the percentage of bottom-of-the-pyramid (BoP) consumers with more adequate diets. The 'Vegetables for All' project has components focused on generating demand for safe and fresh vegetables, improving access to safe and fresh vegetables, and improving the enabling environment to support the policy and regulatory environment within which vegetable value chains function. The project resonates with Uganda's programs and interventions for preventing diet-related non-communicable diseases (DR-NCDs). Further, few evaluations of integrated nutrition and food systems programs have been conducted globally. Therefore, an evaluation of such a program would generate insights that could inform policies and program initiatives for preventing DR-NCDs in Uganda and in other contexts.

Objective: The overall objectives of the evaluation are: 1) To assess the change in the quantity (grams) of vegetables consumed in the last 24 hours before and after GAIN's Vegetables for All Project by women and children 3-9 years in BoP households in the intervention versus control areas in the study districts; 2) To assess the effect of the Vegetables for All project on secondary outcomes in BoP households in intervention versus control areas in study districts; 3) to assess the effect of the Vegetables for All project on knowledge, attitudes, and intentions related to vegetable consumption in BoP households in the intervention versus control areas in study districts; and 4) To conduct a program impact pathway analysis that will provide information that GAIN can use to adapt their program at midline and that will help support the findings of the impact evaluation at endline.

Methods: This evaluation will use a mixed-methods quasi-experimental design in which 136 FFZs are assigned to intervention or control groups across four districts. The impacts will be assessed through cross-sectional population-based surveys of households with women 18-49 years who have a child 3-9 years in the selected FFZs at baseline and endline (N=1,360 at each time point). Vegetable vendor surveys will be conducted in all 136 sampled FFZs at baseline and endline (N=408 at each time point). Qualitative data will be collected at midline and endline. In-depth interviews (IDIs) will be conducted with vegetable value chain actors and other stakeholders (N=16 at midline and endline). Focus group discussions (FGDs) will be conducted with vegetable vendors (16 FGDs at midline and endline) and household members (16 FGDs at midline and endline). The analysis will be performed using difference-in-difference estimation (surveys) and thematic content analysis methods (qualitative). A PIP analysis will be conducted at endline using a combination of qualitative and quantitative data to help understand the pathways through which the program achieved its impact.

ELIGIBILITY:
Different populations will be targeted for different data collection methods. Eligibility criteria are detailed below for each data collection method.

Household Surveys

Inclusion Criteria:

* Reside in the FFZs selected;
* Be a woman between 18-49 years old;
* Have a child 3-9 years old;
* The household earns $250 per month;
* Be able to speak one of the main local languages (Luganda and/or Lusoga);
* Provide informed consent to participate in the study.

Vegetable Vendor Surveys

Inclusion Criteria:

* Be a vegetable vendor in a FFZ in the districts selected for the evaluation;
* Be in business for at least 6 months
* Be over 18 years old;
* Be able to speak one of the main local languages (Luganda and/or Lusoga);
* Provide informed consent to participate in the study.

In-depth interviews with value chain actors:

Inclusion criteria:

* Be a vegetable supplier to vegetable vendors as part of the FFZ, involved in demand generation activities, or involved in food safety compliance;
* Be over 18 years old;
* Be able to speak one of the main local languages (Luganda and/or Lusoga);
* Provide informed consent to participate in the study.

FGDs with vegetable vendors:

Inclusion criteria:

* Work as a vegetable vendor
* Have been a vegetable vendor for at least 6 months
* Be over 18 years old;
* Be able to speak one of the main local languages (Luganda and/or Lusoga);
* Provide informed consent to participate in the study.

Exclusion Criteria:

• For endline: participants will be excluded if they participated in the midline focus group discussion

FGDs with households:

FGD participants will be selected from lists of participants in the FFZ and household surveys and will be consented again for the FGDs if they meet the following criteria:

Inclusion criteria:

* Be a woman living in a BoP household in a FFZ selected for the evaluation;
* Have ever visited a vegetable vendors' place of business;
* Participated in the baseline survey;
* Be over 18 years old;
* Be able to speak one of the main local languages (Luganda and/or Lusoga);
* Provide informed consent to participate in the study.

Exclusion Criteria:

• For endline: participants will be excluded if they participated in a midline FGD

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4616 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Grams of Vegetables Consumed | Baseline (October 2024), Endline (October 2026) (2 years)
  Change in the mean grams of vegetables consumed during the last 24 hours by women and children 3-9 years old in BoP households in Fit Food Zones

CONTACTS AND LOCATIONS:
Overall Officials: Simon Kasasa, Principal Investigator — Makerere University; Valerie Flax, Principal Investigator — RTI International
Locations (1):
- Makerere University School of Public Health, Kampala, Uganda